CLINICAL TRIAL: NCT04001465
Title: Determining Baseline Respiratory Duty Cycles in Subjects With and Without Airway Hyperresponsiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TiTtot-2019
Record Dates: First submitted 2019-06-11; First posted 2019-06-28 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Airway Hyper Responsiveness
MeSH Terms: conditions — Respiratory Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volumetric methacholine challenge (Active Comparator): Methacholine challenge performed per the volumetric method using an Aerogen Solo vibrating mesh nebulizer
  Interventions: Procedure: Volumetric methacholine challenge unmodified
- Methacholine challenge with spirometer (Active Comparator): Methacholine challenge performed per the volumetric method using an Aerogen Solo vibrating mesh nebulizer fitted with an ultrasonic spirometer
  Interventions: Procedure: Modified volumetric methacholine challenge

INTERVENTIONS:
Procedure: Volumetric methacholine challenge unmodified — Bronchoprovocation challenge performed per volumetric method
  Arms: Volumetric methacholine challenge
Procedure: Modified volumetric methacholine challenge — Bronchoprovocation challenge performed per volumetric method modified to include use of ultrasonic spirometer fitted with vibrating mesh nebulizer
  Arms: Methacholine challenge with spirometer

SUMMARY:
The study investigates the inspiratory duty cycle in subjects with and without airway hyper-responsiveness both at rest and during a bronchoprovocation challenge. The primary goal is to determine an average inspiratory duty cycle for standard use in the calculation of bronchoprovocation test results.

DETAILED DESCRIPTION:
At least fifteen subjects with airway hyper-responsiveness and fifteen without airway hyper-responsiveness will be recruited to participate in this randomized, crossover study. Subjects will complete 2 methacholine challenges at least 24 hours apart. One methacholine challenge will entail the volumetric method using a vibrating mesh nebulizer. The second methacholine challenge will be performed identically except that the nebulizer will be fitted onto an ultrasonic nebulizer so as to measure the inspiratory duty cycle throughout the bronchoprovocation challenge.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Participants with airway hyper-responsiveness must have a positive methacholine challenge
* Forced expiratory volume (FEV1) of at least 65% of predicted (based on age, height, and gender)
* Participants without airway hyper-responsiveness must have a negative methacholine challenge
* All participants must avoid strenuous exercise on test days
* No short-acting beta-2 agonist use within 6 hours of study visit

Exclusion Criteria:

* Participants without known airway hyper-responsiveness cannot have a current or historical respiratory condition (e.g. asthma, allergic rhinitis)
* Participants cannot be taking long-acting bronchodilators
* Participants cannot be pregnant or lactating
* Participants cannot have cardiovascular problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Average inspiratory duty cycle in subjects with airway hyper-responsiveness measured using ultrasonic spirometer and tidal breathing | 24 hours
  The inspiratory duty cycles measured for each participant (in duplicate over at least 24 hours) will be averaged for all participants with airway hyper-responsiveness and for all participants without airway-hyperresponsiveness
Average inspiratory duty cycle in subjects without airway hyper-responsiveness | 24 hours
  The inspiratory duty cycles measured for each participant (in duplicate over at least 24 hours) will be averaged for all participants without airway hyper-responsiveness

SECONDARY OUTCOMES:
Within-subject variability in inspiratory duty cycle measured using ultrasonic spirometer and tidal breathing during room air inhalation | 24 hours
  Repeat measurements of inspiratory duty cycle during tidal breathing of room air collected at least 24 hours apart
Between-subject variability within subject group (i.e. airway hyper-responsiveness group) | 1 hour
  Investigation of whether subjects differ in their inspiratory duty cycles (within their respective study group)
Variability in inspiratory duty cycle within subjects when inhaling room air versus an aerosol while using tidal breathing through an ultrasonic spirometer | 1 hour
  Investigation of whether participants differ in their inspiratory duty cycle when inhaling room air versus a saline vapor (i.e. does an aerosol influence people's breathing pattern)
Within-subject variability in provocative dose of methacholine causing a 20% fall in forced expiratory volume (PD20) between repeat methacholine challenges | 24 hours
  Repeat PD20 measures collected for each participant will be compared to determine if there is any significant within-subject variability in PD20
Variability in inspiratory duty cycle with progressive airway constriction induced through methacholine challenge testing | 24 hours
  The inspiratory duty cycle in each subject will be measured throughout a methacholine challenge during each inhalation period, which will allow for determination of whether the inspiratory duty cycle changes with the progressive airway constriction (or lack thereof) induced through methacholine challenge testing
Variability in in inspiratory duty cycle between airway hyper-responsiveness group and group without airway-hyperresponsiveness | 1 hour
  Analysis of variance to determine whether subjects differ in their inspiratory duty cycles based on their status as having or as not having airway-hyperresponsiveness
Within-subject variability in inspiratory duty cycle measured using ultrasonic spirometer and tidal breathing during saline inhalation | 24 hours
  Repeat measurements of inspiratory duty cycle during tidal breathing of nebulized saline collected at least 24 hours apart
Between-subject variability within subject group (no airway hyper-responsiveness group) | 1 hour
  Investigation of whether subjects differ in their inspiratory duty cycles (within their respective study group)

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No